CLINICAL TRIAL: NCT00792532
Title: Use of Interventional MRI for Implantation of Deep Brain Stimulator Electrodes
Acronym: iMRI
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: MRI Interventions, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: iMRI
Record Dates: First submitted 2008-11-14; First posted 2008-11-18 (Estimated); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Parkinson's Disease; Dystonia
MeSH Terms: conditions — Parkinson Disease; Dystonia | interventions — Magnetic Resonance Imaging, Interventional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- iMRI
  Interventions: Procedure: interventional MRI for implantation of DBS electrodes; Device: DBS electrodes

INTERVENTIONS:
Procedure: interventional MRI for implantation of DBS electrodes — DBS implantation will be performed entirely within a Phillips 3T MRI scanner
  Other Names: interventional MR
Device: DBS electrodes — Deep brain stimulation (DBS) electrodes

SUMMARY:
The purpose of this study is to gather observational data on an already FDA-approved implantation technique for deep brain stimulation (DBS) in which the entire surgery is performed within an MRI scanner ("interventional MRI", or iMRI). With this surgical technique, the patient is fully asleep (under general anesthesia) during DBS implantation. The standard method for the placement of deep brain stimulators does not use MRI during the actual DBS placement. The standard method involves placement of a rigid frame on the patient's head, performance of a short MRI scan, transport to the operating room, placement of the DBS electrodes in the operating room, and return to the MRI suite for another MR to confirm correct electrode placement. In the standard method, the patient must be awake for 2-4 hours in the operating room to have "brain mapping" performed, where the brain target is confirmed by passing "microelectrodes" (thin wires) into the brain to record its electrical activity. In the standard method, general anesthesia is not required. With the iMRI technique, the surgery is guided entirely by MRI images performed multiple times as the DBS electrode is advanced. This eliminates the need for the patient to be awake, and eliminates the need for passing microelectrodes into the brain before placing the permanent DBS electrode.

DETAILED DESCRIPTION:
Deep brain stimulation (DBS) is an increasingly common surgical technique for the treatment of Parkinson's disease and dystonia. The current technical approach to DBS implantation involves frame-based stereotaxy. In this method, a stereotactic frame is rigidly fixed to the patient's skull, an MRI is obtained, an anatomic target is identified, and the coordinates of the target in stereotactic space are calculated. Instruments are mounted on the stereotactic frame that point to the calculated coordinate. However, due to the inherent inaccuracies in standard frame-based stereotaxy, a complex 6-hour procedure then ensues to "map" the brain target with microelectrodes, place the lead, and return to the MR unit to confirm proper placement.

The goal of this project is to gather observational data on the iMRI DBS implantation technique and clinical outcomes. This already FDA-approved implantation technique for DBS will take place entirely within the Phillips 1.5T and a Siemens 3T open magnet MRI machine. Prior to study initiation, instrumentation and MR protocols were tested using a phantom head. In the proposed project, subthalamic nucleus or globus pallidus DBS implantations will be performed bilaterally in patients with Parkinson's disease or dystonia. Patients will be under general anesthesia. Targeting and lead verification are performed with imaging alone, without physiologic mapping. Data is to be gathered on the following: operative time, degree of benefit with bilateral implantation (changes in standard rating scales of motor disability), DBS voltage requirements, complications), and electrode location by MR. These measures will be compared with our historical controls, previously entered into our research database, in which electrodes were placed by the standard methods. We expect that the use of near real time MR will improve the speed and accuracy of DBS implantation, and eliminate the need for invasive physiological monitoring.

All of the study participants will be getting iMRI DBS implantation as a part of their standard of care and agree to have additional study data collected

ELIGIBILITY:
Parkinson's Disease

Inclusion Criteria:

1. Diagnosis of idiopathic PD with clinically significant motor fluctuations despite maximized anti-Parkinsonian therapy. This will be based on medical history, neurologic examination (the presence of at least 2 of the following: resting tremor, rigidity, or bradykinesia), and response to anti-Parkinsonian therapy.
2. Approximately 5 years' duration, relative to the date of surgery, since diagnosis of PD.
3. Age >20 inclusive, on date of surgery.
4. The subject is ambulatory in their best on time (not wheelchair bound).
5. The subject is medically able to undergo the surgery as determined by clinical and laboratory evaluations and any other evaluations that are part of the standard practice at the institution in which the subject is to undergo surgery (e.g., subjects will have normal coagulation tests and normal platelet levels).
6. The subject is expected to be able to comply with and understand the required visit schedule and all required tests and procedures.
7. Signed IRB-approved informed consent is obtained before any study-specific procedure, including assessments required during the eligibility evaluation period.

Exclusion Criteria:

1. In the judgment of the investigator, a history of any clinically significant medical, psychiatric, or laboratory abnormality for which participation in the study would pose a safety risk to the subject.
2. History of treatment of PD by any procedure involving intracranial surgery or implantation of a device.
3. MRI of the brain within 12 months before the surgery which demonstrates an intracranial abnormality that would contraindicate surgery (e.g. stroke, tumor, vascular abnormality affecting the DBS target area).
4. Any disorder that precludes a surgical procedure (e.g., signs of sepsis or inadequately treated infection) or alters wound healing.
5. Receipt of antiplatelet agents for at least 10 days prior surgery.
6. Significant cognitive impairment based on investigator assessment during the eligibility evaluation period.
7. History of significant psychiatric illness, epilepsy, or Alzheimer's disease.
8. Active drug or alcohol abuse.
9. Pregnancy or lack of effective contraception in women of childbearing potential defined as one year post-menopausal or surgically sterile.
10. Treatment with non anti-Parkinsonian agents (e.g., atypical neuroleptics) that may affect symptoms of PD within 60 days before entering the study.
11. Any medical disability (e.g., severe degenerative arthritis, compromised nutritional state, severe peripheral neuropathy) that would interfere with the assessment of safety and efficacy in this trial.
12. Inability to follow-up with post-operative study visits
13. Inability to speak or read English

Dystonia Inclusion Criteria

1. Dystonia diagnosed by a movement disorders neurologist
2. Significant functional impairment despite optimal medical management, including failed botulinum toxin therapy if appropriate
3. Age >20 years inclusive, on date of surgery.
4. The subject is medically able to undergo the surgery as determined by clinical and laboratory evaluations and any other evaluations that are part of the standard practice at the institution in which the subject is to undergo surgery (e.g., subjects will have normal coagulation tests and normal platelet levels).
5. The subject is able to comply with and understand the required visit schedule and all required tests and procedures.
6. Signed IRB-approved informed consent is obtained before any study-specific procedure, including assessments required during the eligibility evaluation period.

Exclusion Criteria

1. Any disorder that precludes a surgical procedure (e.g., signs of sepsis or inadequately treated infection) or alters wound healing.
2. Receipt of antiplatelet agents for at least 10 days prior surgery.
3. Significant cognitive impairment based on investigator assessment during the eligibility evaluation period.
4. History of significant psychiatric illness, epilepsy, or Alzheimer's disease.
5. Active drug or alcohol abuse.
6. Pregnancy or lack of effective contraception in women of childbearing potential defined as one year post-menopausal or surgically sterile.
7. Any medical disability (e.g., severe degenerative arthritis, compromised nutritional state, severe peripheral neuropathy) that would interfere with the assessment of safety and efficacy in this trial.
8. Inability to follow-up with post-operative study visits
9. Inability to speak or read English

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson's disease, eligible for DBS
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2003-07 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Parkinson's disease: The degree of benefit from baseline off medication UPDRS(part III) motor score to postoperative off medication scores at 12 months with stimulation on. | 12 months post-surgery
Dystonia: The percent change from baseline in the Burk-Fahn-Marsden Dystonia rating scale movement subscore to the 12 month postoperative subscore | 12 months post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Philip Starr, M.D., Ph.D., Principal Investigator — University of California, San Francisco; SFVAMC; Paul Larson, M.D., Principal Investigator — University of California, San Francisco; SFVAMC; Jill L Ostrem, MD, Principal Investigator — University of California San Francisco, SFVAMC; Alastair J Martin, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco VA Medical Center, San Francisco, California, United States

REFERENCES:
- [Result] Martin AJ, Larson PS, Ostrem JL, Keith Sootsman W, Talke P, Weber OM, Levesque N, Myers J, Starr PA. Placement of deep brain stimulator electrodes using real-time high-field interventional magnetic resonance imaging. Magn Reson Med. 2005 Nov;54(5):1107-14. doi: 10.1002/mrm.20675. PMID 16206144
- [Derived] Ostrem JL, Ziman N, Galifianakis NB, Starr PA, Luciano MS, Katz M, Racine CA, Martin AJ, Markun LC, Larson PS. Clinical outcomes using ClearPoint interventional MRI for deep brain stimulation lead placement in Parkinson's disease. J Neurosurg. 2016 Apr;124(4):908-16. doi: 10.3171/2015.4.JNS15173. Epub 2015 Oct 23. PMID 26495947
- [Derived] Starr PA, Markun LC, Larson PS, Volz MM, Martin AJ, Ostrem JL. Interventional MRI-guided deep brain stimulation in pediatric dystonia: first experience with the ClearPoint system. J Neurosurg Pediatr. 2014 Oct;14(4):400-8. doi: 10.3171/2014.6.PEDS13605. Epub 2014 Aug 1. PMID 25084088